CLINICAL TRIAL: NCT06426381
Title: The Effect of Therapeutic Touch Applied During Knee Replacement Surgery on Anxiety, Vital Signs and Comfort Level / Experimental Randomized Controlled Trial
Brief Title: The Effect of Therapeutic Touch Applied During Knee Replacement Surgery on Anxiety, Vital Signs and Comfort Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilek GÜRÇAYIR (Other)
Responsible Party: Sponsor-Investigator, Dilek GÜRÇAYIR, Academician, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ayse25
Record Dates: First submitted 2024-05-07; First posted 2024-05-23 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Intraoperative Complications
Keywords: therapeutic touch; anxiety; comfort
MeSH Terms: conditions — Intraoperative Complications; Anxiety Disorders | interventions — Therapeutic Touch

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- There is therapeutic touch (Experimental): Patients will be administered an Introduction Form and Spielberg State-Trait Anxiety Scale before surgery. The Vital Signs Record Form will be filled out on the patient's operating table. Then, therapeutic touch will be applied for 15-20 minutes during the surgery. After the procedure, the Vital Signs Record Form, Spielberg State Anxiety Scale and Perianesthesia Comfort Scale (PCS) will be administered.
  Interventions: Behavioral: Therapeutic Touch
- No therapeutic touch (No Intervention): An Introduction Form and the Spielberg State-Trait Anxiety Scale will be administered to the patients. When you are taken to the operating table, a Vital Signs Record Form will be filled out. After the procedure is completed, the Vital Signs Record Form, Spielberg State Anxiety Scale and Perianesthesia Comfort Scale (PCS) will be administered.

INTERVENTIONS:
Behavioral: Therapeutic Touch — Asymmetric energy fields can be balanced using the therapeutic touch method and treatment becomes easier. In this way, the person regains his health or can be helped to regain his health.
  Arms: There is therapeutic touch

SUMMARY:
The aim of this study is to investigate the effect of therapeutic touch on patients' anxiety, vital signs and comfort levels during knee replacement surgery performed under local anesthesia.

The study will be completed with a total of 128 participants, including 64 experimental and 64 control participants.

As a randomization method, the simple randomization method will be used to ensure an equal number of samples in two groups, and patients will be assigned to the experimental and control groups. In the research, patients will be given verbal information about the research, and written informed consent will be obtained from the patients who accept it.

In the study, therapeutic touch was applied for 15-20 minutes during knee replacement surgery and the effect of this application on vital signs, anxiety level and comfort was evaluated.

DETAILED DESCRIPTION:
Knee replacement surgeries are a common treatment method for patients with problems such as pain and limitation of movement resulting from knee joint disorders. This type of surgery is usually performed under general anesthesia, allowing patients to lose consciousness during surgery. However, general anesthesia may have some risks and complications. For this reason, local anesthesia has become increasingly popular.

Local anesthesia is a method of anesthesia used to numb the surgical area. In this method, anesthesia is injected directly into the surgical area and the patient is awake and conscious throughout the surgery. Local anesthesia may have fewer side effects and complications compared to general anesthesia. However, the effects of emotional factors such as stress, anxiety and discomfort experienced by patients during surgeries performed under local anesthesia are still poorly understood .

The human body is surrounded by an aura and open energy fields. It is reported that when these energy fields are balanced, the individual is healthy, and when they are irregular, the individual experiences health problems. Asymmetric energy fields can be balanced using the therapeutic touch method and treatment becomes easier. In this way, the person regains his health or can be helped to regain his health. Nursing theorist Martha Rogers supports this statement. Rogers defined human beings as an open system with a complex and interactive energy field covering the entire universe. It is assumed that the energy surrounding humans is in wave form and that changes in the human body are controlled by these energy fluctuations. If the person has health problems, this manifests itself in the form of energy blockages or rhythm disorders. By correcting these energy rhythm disorders discovered by the nurse with the therapeutic touch method, the person's health problem can be treated. In recent years, there has been increasing evidence that alternative approaches, such as therapeutic touch, have positive effects on surgical outcomes. Therapeutic touch is a method that aims to provide relaxation, calming and healing through physical contact. This method can reduce patients' stress levels, relieve pain, and increase their overall comfort level. However, there are limited studies on the effect of therapeutic touch on vital signs during knee replacement surgery performed under local anesthesia.

Surgeries are widely used as a method of treating various health problems that require medical treatment. Knee prosthesis surgeries are one of the frequently used surgical interventions in the treatment of painful and limiting diseases of the knee joint. Although such surgeries have the potential to significantly improve individuals' mobility and quality of life, the stress, anxiety and physical discomfort that may occur during and after the surgery can be a significant source of concern for patients.

Anxiety is a common psychological reaction before and after surgical interventions and is an important factor affecting the surgical process. Patients may experience increased levels of anxiety when faced with uncertainty about the results of surgery, possible complications, and the recovery process. The importance of this situation is of great importance in terms of the success of the surgery and the patients' ability to better manage the postoperative period.

Anxiety negatively affects the patient's comfort level after surgery and can prolong the recovery process. Lack of comfort can lead to increased physical and emotional stress caused by surgery. It is important to note that because therapeutic touch has the potential to increase patients' relaxation, stress reduction, and overall comfort level, research has also been conducted in this area. However, there is no definitive information about the effect of therapeutic touch on the comfort level during knee replacement surgery performed under local anesthesia.

The aim of this study is to investigate the effect of therapeutic touch on patients' vital signs, anxiety and comfort level during knee replacement surgery performed under local anesthesia. This study aims to offer an alternative approach to improve patients' quality of life by continuing to improve the results of surgeries performed under local anesthesia. This study aims to fill the gap in this field by investigating the effect of therapeutic touch on vital signs, anxiety and comfort level during knee replacement surgery performed under local anesthesia. The findings may guide clinical practice in providing an alternative approach to improve surgical outcomes and reduce discomfort experienced by patients. It may also provide basic information to evaluate the feasibility of therapeutic touch in other surgical procedures under local anesthesia.

This study was conducted as an experimental randomized controlled study. This method was preferred because it allows the situations and attitudes of the individuals in the group selected as a sample, regarding a phenomenon or event, and to describe the phenomena and events in their own conditions and as they are. In addition, in randomized controlled studies, the factors that cause events and situations and the degree of influence of these factors can be determined. In the study, therapeutic touch was applied for 15-20 minutes during knee replacement surgery and the effect of this application on vital signs, anxiety level and comfort was evaluated. The hypotheses created in the research are listed below; The research was conducted in the orthopedics and traumatology room in the operating room department of Atatürk University Training and Research Hospital between September 2023 and June 2024.

The population of the research consists of patients who had knee replacement surgery between September 2023 and February 2024. The sample of the research consists of patients who meet the inclusion criteria between the specified dates. Cohen's standard effect sizes were used as reference in the power analysis. In this case, in this study, for the t test in independent groups where the effect of therapeutic touch during knee prosthesis surgery will be compared on vital signs, anxiety and comfort levels, if the study is conducted with a total of 128 participants in two groups with 64 participants in each group, 80% confidence interval is 95% at a significance level of 0.05. It has been determined that power can be achieved. As a randomization method, the "simple randomization method" was used to ensure an equal number of samples in two groups, and the patients were assigned to the experimental and control groups. In the study, patients were given verbal information about the research, and written informed consent was obtained from the patients who agreed.

Four different forms were used to collect data in the study. The Anxiety and Comfort Scale, which was determined as the data collection tool in the study, was chosen by the researcher as it was deemed suitable for the purpose. Analyzes were carried out with the data obtained to test the validity and reliability of the selected scale. In order to ensure that the data collection tools do not pose an ethical problem, people with expertise on the subject were consulted and it was ensured that they would not cause any problems. However, the scale questions were reviewed in detail by the researcher and the consultant, and since an application was actually made in the form of a Likert scale, leaving the selection decision entirely to the participants refutes the idea that it is a manipulation. The forms used to collect data are listed below;

1. Patient Introduction Form
2. Vital Signs Record Form
3. Spielberg State-Trait Anxiety Scale
4. Perianesthesia Comfort Scale (PCS) In order to conduct the research, firstly, approval was obtained from the Atatürk University Faculty of Medicine Ethics Committee and institutional permission was obtained from the hospital where the research was conducted. Verbal consent was obtained from the patients before data collection, and data collection forms were collected by the researcher in the orthopedics and traumatology room in the operating room department by face-to-face interview. Patients who accepted the study and met the criteria were included in the experimental/control group by randomization.

In patients included in the experimental group; On the day of surgery, patients who met the research criteria were met, the purpose of the study was explained, and their written consent was obtained. The Patient Introduction Form and the Spielberg State-Trait Anxiety Scale were administered in the patient room using face-to-face interview technique. When the patient was taken to the operating table, the Vital Signs Record Form was filled out. Then, therapeutic touch was applied for 15-20 minutes during the surgery. After the procedure was completed, the Vital Signs Record Form, Spielberg State Anxiety Scale and Perianesthesia Comfort Scale (PCS) were administered.

In patients included in the control group; On the day of surgery, patients who met the research criteria were met, the purpose of the study was explained, and their written consent was obtained. The Patient Introduction Form and the Spielberg State-Trait Anxiety Scale were administered in the patient room using face-to-face interview technique. When the patient was taken to the operating table, the Vital Signs Record Form was filled out. After the procedure is completed, the Vital Signs Record Form, Spielberg State Anxiety Scale and Perianesthesia Comfort Scale (PCS) will be administered. No procedure was applied to the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 18-85
2. No communication problems (speaks Turkish)
3. No vision or hearing problems
4. No cognitive problems
5. The patient agrees to participate in the study
6. Having knee replacement surgery with local anesthesia

Exclusion Criteria:

1. Being under the age of 18 and over the age of 85
2. Having a communication problem (does not speak Turkish)
3. The patient wants to leave the study
4. Not agreeing to participate in the research
5. Not being at a cognitive level to answer the questions asked.
6. Patients with vision and hearing problems
7. Having knee replacement surgery with general anesthesia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Patient Introduction Form | up to 24 weeks
  The survey form, created by the researcher by scanning the literature on the subject, consists of a total of 13 questions including questions about gender, age, place of residence, education, status, profession, marital status, and total knee replacement surgery.
Vital Signs Record Form | up to 24 weeks
  An observation form was used to observe the patients in the experimental and control groups to whom therapeutic touch was applied during surgery. This form was used to record the duration of therapeutic touch, respiration, oxygen saturation, pulse, systolic blood pressure, and diastolic blood pressure.
Spielberg State-Trait Anxiety Scale | Before and after surgery
  There are 4 different options in the section that the individuals to whom the scale is applied will mark. These options consist of "not at all", "somewhat", "a lot" and "completely" in order to determine the intensity of the expressed behaviors and emotions. The total score obtained from both scales varies between 20-80. High scores indicate high anxiety levels, low scores indicate low anxiety levels. There are two types of statements in the State-Trait Anxiety Scale. Direct expressions express negative emotions, while inverted expressions express positive emotions. The reversed expressions in the State Anxiety Scale are items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20. The reversed expressions in the Trait Anxiety Scale constitute items 26, 27, 30, 33, 36 and 39. After finding the total weights of direct and reverse expressions separately, the total weight score of reverse expressions is subtracted from the total weight score obtained for direct expressions.
Perianesthesia Comfort Scale (PCS) | up to 24 weeks
  The scale consists of 24 items that reflect the individual's general thought process before and after the surgical intervention and question his/her self-conception and feelings. Each statement in the scale has a Likert-type scoring ranging from 1 to 6, from "strongly disagree" to "strongly agree". The response patterns of the scale, which consists of positive and negative items, are given in mixed order. 12 of the statements are positive (1.5, 6, 11, 14, 16, 18, 19, 20, 21, 23, 24), 12 are negative (2, 3, 4, 7, 8, 9, 10, 12, 13, 15, 17, 22); Negative statements are reversed in scoring. Accordingly, in positive statements, a high score (6) indicates high comfort, a low score (1) indicates low comfort, and in negative items, a low score (1) indicates high comfort and a high score (6) indicates low comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek GÜRÇAYIR, Dr., Principal Investigator — Ataturk University
Locations (1):
- Ayşe ÇELİK, Palandöken, Erzurum, Turkey (Türkiye)